CLINICAL TRIAL: NCT06748118
Title: Improving Patients' Adherence to Their Chronic Treatments by Implementing a Simple, Standardized and Redundant Message Delivered by Healthcare Professionals: a Stepped-wedge Multicenter Randomized Trial
Brief Title: Improving Patients' Adherence to Their Chronic Treatments by Implementing a Simple, Standardized and Redundant Message Delivered by Healthcare Professionals.
Acronym: MAPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: APHP230810; PREPS-22-0004 (Other Grant/Funding Number: French Ministry of Health); DR-2024-271 (Other: Commission Nationale de l'Informatique et des Libertés); 2024-A00701-46 (Other: ANSM)
Record Dates: First submitted 2024-12-05; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: Chronic Disease; Therapeutic Adherence; Training Group, Sensitivity; Delivery Simple, Standardized & Redundant Message to Patient
Keywords: intervention study; stepped wedge study
MeSH Terms: conditions — Chronic Disease; Treatment Adherence and Compliance; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: The research is multicentric and randomized. The study intervention will be implemented in a stepped-wedge design with 10 steps, 10 healthcare facilities (clusters), 12 2-month periods, 1 2-month period including wash-out and training of healthcare professionals (intervention). The wash-out will prevent contamination between the two periods.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention period (Experimental): Trained healthcare professionals deliver a simple, standardized and redundant 3-point message to patients, based on the levers of action for therapeutic adherence.
  During this period, the message will be delivered to the patient by each of the healthcare professionals involved in his or her hospital care. It will be formalized by a checklist that will enable them to reformulate the 3 points defined as key elements of therapeutic adherence. Each healthcare professional is free to deliver this message at any time during their consultation/interview with the patient. They will be asked to note the date and tick off each point on the checklist.
  The intervention period will take place after the control and wash-out periods, and after healthcare professionals have been trained in the intervention.
  Interventions: Other: Trained healthcare professionals deliver a simple, standardized and redundant 3-point message to patients, based on the levers of action for therapeutic adherence.
- Control period (No Intervention): The control period is the period before healthcare professionals are trained in the intervention. Patients included during this period will not receive the simple, standardized and redundant message.

INTERVENTIONS:
Other: Trained healthcare professionals deliver a simple, standardized and redundant 3-point message to patients, based on the levers of action for therapeutic adherence. — This message is delivered with the aim of modifying the patient's behavior with regard to treatment intake. The research does not anticipate any change in the patient's medical prescriptions.
  Other Names: Intervention period
  Arms: Intervention period

SUMMARY:
The primary objective in this study is to achieve a 15% 6-month improvement in therapeutic adherence among patients with chronic pathologies, thanks to a simple, standardized and redundant message delivered by healthcare professionals during consultations/interviews Trained healthcare professionals deliver a simple, standardized and redundant 3-point message to patients, based on the levers of action concerning therapeutic adherence. This message is delivered with the aim of modifying the patient's behavior with regard to treatment intake.

DETAILED DESCRIPTION:
This project will enable us to adapt or even modify the practices of healthcare professionals, by making management recommendations to improve patients' adherence to treatment during their consultations/interviews, and throughout their entire course of care. This project will increase the benefit/risk ratio of treatments and reduce the waste of healthcare resources.

For patients, their participation by filling in the therapeutic adherence self-questionnaire will enable them to become active players in the management of their treatment.

If the results of our study prove positive, this will lead to a new, optimized organization of patient care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years)
* Affiliated to the French social security system
* Followed in hospital for a chronic pathology within a formalized care pathway
* Having signed a consent form to participate in the study.

Exclusion Criteria:

* Patients included in the control period.
* Patients under guardianship.
* Pregnant or breast-feeding patients.
* Patients taking part in research on compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1210 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Improvement in therapeutic adherence | 6 months
  The medication possession ratio (MPR), calculated as the ratio between the sum of treatment days delivered over the period of interest x 100, expressed as a %. In the literature, an MPR ≥ 80% corresponds to good therapeutic adherence.

SECONDARY OUTCOMES:
Improvement in therapeutic adherence | 12 months
  The medication possession ratio (MPR), calculated as the ratio between the sum of treatment days delivered over the period of interest x 100, expressed as a %.
Predictive factors of improved adherence factors predictive of therapeutic adherence | 6 months
  Identification of predictive factors for improving adherence assessed by the Freedom patient self-questionnaire and known factors.
Improvement in therapeutic adherence estimated | 12 months
  patient adherence self-questionnaire, taking into account what the patient says between M0 and M3, M3 and M6; and between M0 and M12, M6 and M12 (11 questions formulated using a 5-point Likert scale), which classifies patients' therapeutic adherence into 3 classes: "low therapeutic adherence / average / high". Improvement in adherence will be assessed by changing the adherence category.
Costs of care according to periods (control vs. intervention) | 12 months
  The number of consultations (general practitioner, specialist, nurse), hospital admissions (day and conventional), emergency room visits, and the number and duration of days off work will be collected prospectively via a questionnaire on the evaluation of healthcare use given to the patient at M0, M3, M6 and M12. Costs will then be evaluated using the official tariffs for each procedure or hospitalization. Treatment costs will be evaluated on the basis of data from copies of prescriptions collected by pharmacists at each center.
Cost of the intervention | 12 months
  a comparison of the cost of the intervention in terms of time spent on training by healthcare professionals and delivery of the 3-point message for each patient will be carried out, compared with the control group.
Satisfaction of participating healthcare professionals and reasons for refusal to participate | 12 months
  Numbers and percentages will be reported for each question of the professional satisfaction self-questionnaire adapted from Jean-Marc Palm questionnaire. The questionnaire contains six questions. The answers range from totally disagree to totally agree.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte SABATIER, Dr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (10):
- France (10):
  - CHU d'Angers, Angers, France
  - CH d'Antibes, Antibes, France
  - Hôpital Corentin Celton, Issy-les-Moulineaux, France
  - Hôpital de la Conception, Marseille, France
  - Hôpital La Timone, Marseille, France
  - CHU de Nantes, Nantes, France
  - Hôpital européen Georges-Pompidou, Paris, France
  - Hôpital Bicêtre, Paris, France
  - CHU de Toulouse, Toulouse, France
  - CHU de Tours, Tours, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. The founder could be involved in the decision. Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization. Processing of shared data must comply with European General Data Protection Regulation (GDPR).